CLINICAL TRIAL: NCT01044004
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study to Evaluate the Efficacy of Armodafinil for Patients With B-cell Lymphoma and Severe Fatigue Undergoing Standard R-CHOP Chemotherapy or in Remission Following Chemo and/or Radiation
Brief Title: Evaluate the Efficacy of Armodafinil for Patients With B-cell Lymphoma and Severe Fatigue
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 09-1896
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: B-cell Lymphoma; Fatigue
MeSH Terms: conditions — Lymphoma, B-Cell; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Post treatment remission armodafinil (Experimental): Armodafinil 150 mg/day for 13 weeks
  Interventions: Drug: Armodafinil
- Post treatment remission placebo (Placebo Comparator): Placebo 150mg/day for 13 weeks
  Interventions: Drug: placebo
- Chemotherapy armodafinil (Experimental): Armodafinil 150 mg/day for 13 weeks
  Interventions: Drug: Armodafinil
- Chemotherapy placebo (Placebo Comparator): Placebo 150mg/day for 13 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Armodafinil — Armodafinil 150 mg/day for 13 weeks
  Other Names: Nuvigil
  Arms: Post treatment remission armodafinil
Drug: placebo — Placebo 150mg/day for 13 weeks
  Arms: Post treatment remission placebo
Drug: Armodafinil — Armodafinil 150 mg/day for 13 weeks
  Other Names: Nuvigil
  Arms: Chemotherapy armodafinil
Drug: placebo — Placebo 150mg/day for 13 weeks
  Arms: Chemotherapy placebo

SUMMARY:
To determine whether armodafinil is more effective than placebo in reducing fatigue.

DETAILED DESCRIPTION:
Aims will be analyzed separately as stratified by treatment arm (chemotherapy treatment arm vs. post-treatment remission arm).

Primary Objective:

* To determine whether armodafinil is more effective than placebo in reducing fatigue as measured by the change in scores from the FACT-Fatigue reported at study entry, week 7 of study treatment, and study completion (week 13).

Secondary Objectives:

* To determine whether armodafinil is more effective than placebo in reducing fatigue as measured by standard actigraphy summary statistics including total sleep time (TST), wake after sleep onset (WASO), sleep latency, number of awakenings, daytime sleep time, mean daytime activity, peak activity, acrophase, and circadian mesor at week 1 of screening, week 7 of study treatment, and study completion (week 13).
* To determine whether armodafinil is more effective than placebo in improving work quality as measured by the change in scores from the WLQ© reported at study entry (week 1) and study completion (week 13).
* To determine whether armodafinil is more effective than placebo in reducing fatigue as measured by the change in activity patterns with actigraphy using applied functional data analysis during week 1 of screening, week 7 of study treatment, and study completion (week 13).
* To evaluate whether measured cytokines (IL-2, IL-6, IL-10, TNF-α, and TGF-α) are elevated at baseline.
* To evaluate whether measured cytokines (IL-2, IL-6, IL-10, TNF-α, and TGF-α) change from the time of study entry to study completion.
* To assess whether cytokine levels (IL-2, IL-6, IL-10, TNF-α, and TGF-α) correlate with circadian patterns in wrist actigraphy and self-described reports of fatigue as measured by the FACT-Fatigue at baseline and study completion.

ELIGIBILITY:
Inclusion Criteria for both arms:

* Age ≥ 18 with diagnosis of B-cell lymphoma
* Average score of ≥ 7 on daily worst fatigue severity assessment from the BFI questionnaire during screening
* Able to demonstrate appropriate use of the wrist actigraphy device and to complete questionnaires
* ECOG performance status 0-2
* Laboratory values:
* Hemoglobin ≥ 10 g/dL
* Total Bilirubin ≤ 1.5 x institutional ULN
* AST/ALT ≤ 2.5 x institutional ULN
* Creatinine ≤ 1.5 x institutional ULN
* Albumin ≥ 3.5 g/dl
* Life expectancy > 6 months
* IRB-approved informed consent form must be signed before any protocol-specific screening procedures are performed.

Inclusion criteria for patients undergoing R-CHOP chemotherapy:

* Scheduled to receive 6 cycles of standard R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) chemotherapy as first-line treatment

Inclusion criteria for patients in remission following chemotherapy and/or radiotherapy:

* May have received one prior regimen of chemotherapy and/or radiotherapy
* Adequate response to upfront chemotherapy and/or radiotherapy
* Indolent lymphomas - must have achieved a partial or complete response with no immediate plans for further treatment
* Aggressive lymphomas - must have achieved a complete response:

  * ≥ 4 weeks since completion of chemotherapy
  * ≥ 8 weeks since completion of radiotherapy
  * ≤ 18 months since completion of chemotherapy or radiotherapy

Exclusion Criteria for both arms:

* Uncontrolled medical and/or psychiatric condition that may cause fatigue or that the PI feels is clinically significant and might adversely affect patient safety (such as sleep disorders, moderate/severe depression, metabolic/endocrine abnormalities, infections)
* History of clinically significant cardiac disorders, such as left ventricular hypertrophy or mitral valve prolapse experienced in conjunction with receiving CNS stimulants
* History of serious skin reactions, such as serious rash or Stevens-Johnson Syndrome
* Concurrent stimulant medication
* Any other active malignancy within the past 3 years except cervical carcinoma in situ and non-melanoma skin cancers
* Known CNS involvement by lymphoma
* Cachexia
* Use of opioids at time of randomization
* Known sensitivity to modafinil and/or armodafinil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
To determine whether armodafinil is more effective than placebo in reducing fatigue as measured by the change in scores from the FACT-Fatigue reported at study entry, week 7 of study treatment, and study completion (week 13). | 13 weeks

SECONDARY OUTCOMES:
To determine whether armodafinil is more effective than placebo in improving work quality as measured by the change in scores from the WLQ© reported at study entry (week 1) and study completion (week 13). | 13 weeks
To determine whether armodafinil is more effective than placebo in reducing fatigue as measured by standard actigraphy summary statistics will be done at week 1 of screening, week 7 of study treatment, and study completion (week 13). | 13 weeks
To determine whether armodafinil is more effective than placebo in reducing fatigue as measured by actigraphy using applied functional data analysis during week 1 of screening, week 7 of study treatment, and study completion (week 13). | 13 weeks
To evaluate whether measured cytokines (IL-2, IL-6, IL-10, TNF-α, and TGF-α) are elevated at baseline. | 13 weeks
To evaluate whether measured cytokines (IL-2, IL-6, IL-10, TNF-α, and TGF-α) change from the time of study entry to study completion. | 13 weeks
To assess whether cytokine levels (IL-2, IL-6, IL-10, TNF-α, and TGF-α) correlate with circadian patterns in wrist actigraphy and self-described reports of fatigue as measured by the FACT-Fatigue at baseline and study completion. | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nina Wagner-Johnston, M, Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu